CLINICAL TRIAL: NCT01745315
Title: Comparison of the Use of LigaSure, Halo PKS Cutting Forceps and Enseal Tissue Sealer in Total Laparoscopic Hysterectomy: a Randomised Trial.
Brief Title: Comparison of Perioperative Outcomes of Three Different Instruments in Total Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adana Numune Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hakan Aytan, Associate Professor,, Adana Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: instruments in TLH
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Perioperative Outcomes
Keywords: total laparoscopic hysterectomy; LigaSure; EnSeal; Halo PKS Cutting forceps; electrothermal bipolar vessel sealer; advanced bipolar device

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LigaSure (advanced bipolar device) (Active Comparator): Laparoscopic hysterectomy will be done with LigaSure in 15 patients.
  Interventions: Device: Advanced bipolar devices
- Halo PKSforceps(advanced bipolar device) (Active Comparator): Laparoscopic hysterectomy will be done with Halo PKS cutting forceps in 15 patients.
  Interventions: Device: Advanced bipolar devices
- EnSeal (advanced bipolar device) (Active Comparator): Laparoscopic hysterectomy will be done with EnSeal in 15 patients.
  Interventions: Device: Advanced bipolar devices

INTERVENTIONS:
Device: Advanced bipolar devices
  Other Names: LigaSure; Halo PKS cutting forceps; EnSeal

SUMMARY:
There are many instruments with different energy modalities or with different properties that are available for use in total laparoscopic hysterectomy. The aim of the present study is to compare three of these instruments that are present in our clinic - HALO PKS Cutting Forceps, LigaSure and Enseal Tissue Sealer, in total laparoscopic hysterectomy with respect to operation time, blood loss, change in hemoglobin / hematocrit levels, perioperative complications, return of gastrointestinal activity and hospitalization time.

ELIGIBILITY:
Inclusion Criteria:

* any women with the indication of hysterectomy

Exclusion Criteria:

* malignancy
* having 3 or more previous abdominal surgeries
* uterus being larger than 12 weeks of gestation
* patients who must undergo additional surgical procedures during the same operation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Perioperative Outcomes | Until 45 patients are operated (6 months anticipated)
  Perioperative outcomes will be assessed with respect to complication rates, operation time, blood loss, change in hemoglobin and hemotocrit levels, time to return of gastrointestinal function and hospitalization time.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Aytan, M.D., Principal Investigator — Adana Numune Training and Research Hospital
Locations (1):
- Adana Numune Training and Research Hospital, Adana, Turkey (Türkiye)